CLINICAL TRIAL: NCT06266702
Title: Evaluation of a Lipid-based Nutritional Technology for Enhancing Vitamin D Absorption in Humans
Brief Title: Evaluation of a Nutritional Technology for Vitamin D Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: BL71
Record Dates: First submitted 2024-01-08; First posted 2024-02-20 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Nutrition, Healthy
MeSH Terms: interventions — Phospholipids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1A - High Vitamin D, Experimental Oil (Experimental): High dose Vitamin D mixed with Experimental Oil
  Interventions: Other: Experimental Oil with Phospholipids
- Group 1B - High Vitamin D, Control Oil (Active Comparator): High Dose Vitamin D mixed with Control Oil
  Interventions: Other: Control Polyunsaturated Oil Blend
- Group 2A - Low Vitamin D, Experimental Oil (Experimental): Low dose Vitamin D mixed with Experimental Oil
  Interventions: Other: Experimental Oil with Phospholipids
- Group 2B - Low Vitamin D, Control Oil (Active Comparator): Low Dose Vitamin D mixed with Control Oil
  Interventions: Other: Control Polyunsaturated Oil Blend

INTERVENTIONS:
Other: Experimental Oil with Phospholipids — Consumed on white bread
  Arms: Group 1A - High Vitamin D, Experimental Oil; Group 2A - Low Vitamin D, Experimental Oil
Other: Control Polyunsaturated Oil Blend — Consumed on white bread
  Arms: Group 1B - High Vitamin D, Control Oil; Group 2B - Low Vitamin D, Control Oil

SUMMARY:
This is a prospective, 2-group crossover, randomized, double-blind study to evaluate nutrient absorption.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (18-55 years of age)
* Body mass index (BMI) <30 kg/m2
* Males and nonpregnant, nonlactating females
* Free of gastrointestinal disorders that my impact nutrient absorption in the small intestine, endocrine, hepatic, renal, or bone diseases

Exclusion Criteria:

* Use of vitamin D or calcium supplements within 3 weeks prior to the Screening Visit.
* Use of a tanning booth/lamp within 3 weeks prior to the Screening Visit.
* Travel to sunny location within 3 weeks prior to the Screening Visit.
* Consumption of more than 3 alcoholic drinks per day starting 48 hours before the Screening Visit.
* Has an allergy or intolerance to any ingredient in the study product.
* Participating in another study that has not been approved as a concomitant study by Abbott Nutrition.
* Use of the following medications that may have interactions with vitamin D absorption or metabolism:

  * Aluminum-containing phosphate binders
  * Anticonvulsants
  * Atorvastatin
  * Calcipotriene
  * Cholestyramine
  * Cytochrome P-450 3A4 substrates
  * Digoxin
  * Diltiazem
  * Orlistat
  * Thiazide diuretics
  * Corticosteroids
  * Stimulant laxatives
  * Verapamil

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Vitamin D Absorption | Time 0 to 24 Hours
  Change in area under the curve (AUC) of serum vitamin D for low dose in experimental versus control oil

SECONDARY OUTCOMES:
Vitamin D Absorption - Peak | Time 0 to 48 Hours
  Change in Peak serum for vitamin D in experimental versus control oil
Vitamin D Absorption - AUC | Time 0 to 48 Hours
  Change in AUC for vitamin D in experimental versus control oil

OTHER OUTCOMES:
Body Mass Index | Visit 1, Baseline Collection
  As calculated from height in cm and weight in kg
Adverse Events | Study Day 1 to Study Day 7 up to 20 Days
  Participant reported adverse events during study duration

CONTACTS AND LOCATIONS:
Overall Officials: Steve Hertzler, Study Chair — Abbott Nutrition
Locations (1):
- Walsh University, North Canton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No